CLINICAL TRIAL: NCT03319589
Title: Pilot Study on a Locally Prepared Food Supplement to Support Growth and Brain Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: International Partners for Human Development (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200
Record Dates: First submitted 2016-03-11; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition | interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Supplement Arm (Experimental): School children (age 6 to 6.5) will receive their supplement 5 days a week in the morning before school starts. They will either receive the supplement at school or at the community health center depending on the preference of the villagers after recruitment. Young children (age 24 to 30 months) will receive the supplement 5 days a week in the morning at the community health center, distributed by community health workers.
  Interventions: Dietary Supplement: Supplement
- Control Arm (No Intervention): Children in the active intervention village will be compared with assessment-only controls in a separate village having comparable demographic characteristics

INTERVENTIONS:
Dietary Supplement: Supplement — locally prepared biscuit with low sugar content (less than 10% weight) designed to facilitate growth and cognitive development
  Arms: Supplement Arm

SUMMARY:
This study is a randomized controlled pilot for a future larger trial. The goals of this pilot are: a) to assess feasibility of delivering a locally prepared supplement in rural communities, and b) to generate pilot data for sample size estimates needed for a larger trial. The study will test the effect of a supplement prepared locally with local and imported ingredients on changes in standard anthropometric benchmarks of growth, cognition, immune function, hemoglobin and skin carotenoids in young children living in 2 villages in rural Guinea-Bissau. Children in the active intervention village will be compared with assessment-only controls in a separate village having comparable demographic characteristics. As part of the study, we will assess the feasibility of having local commercial bakers prepare the supplement.

DETAILED DESCRIPTION:
Up to 20 children aged 24-30 months and 20 school children aged 6-6.5 years living in each of 2 villages in the Oio region of Guinea-Bissau (total study population up to 80, with no minimum recruitment number) will be recruited for this study, with ages documented by the official birth record, which all families possess. Villages will be a convenience sample chosen from villages within the network of our local research partner International Partnership for Human Development. Each village in this region has one school and one community health center per village, which will be involved in supplement distribution and some outcome assessments. The villages will be broadly comparable in terms of size, affluence, rates of malnutrition, the presence or absence of a school meal program, and tribal affiliation and religion.

One village will be randomly assigned to receive the locally-prepared biscuit and a daily multivitamin and the other will be randomly assigned to be an assessment-only control site. Because this is a pilot study designed to develop methodology for a future powered trial, and the logistics of local supplement preparation need to be developed in advance of the study, the randomization will occur prior to baseline testing to allow for development of infrastructure for supplement preparation. However the villagers will not be informed of the randomization until after baseline testing is complete.

Following baseline measurements of anthropometry, grip strength, cognition, non-invasive measurements of hemoglobin, and skin carotenoids, participants will receive their intervention for 12 weeks and the same measurements taken at baseline will be repeated during the last study week. Since access for the final assessment to villages may be hampered by the rainy season we also request permission to terminate the trial between 9-12 weeks of supplement consumption depending on weather conditions. Please note that cell phone access to villages is not influenced by local weather, thus communication regarding safety issues with community health workers will remain possible throughout the entire trial.

ELIGIBILITY:
Inclusion Criteria:

* Non-malnourished children within the 2 villages chosen for study
* Within the specified age range: 24-36 months for young children and 6-7 years for older children, who will also be enrolled in their local school. In the event that researchers cannot enroll at least 15 participants in each age range in each village, will extend the age range up to 35.99 months for young children and up to 6.99 years for older children.
* The family plans to remain in the village for the duration of the study;
* The child does not have any known food allergies as reported by the mother or guardian.

Exclusion Criteria:

* If any child is identified as malnourished at baseline, defined as a mid-upper arm circumference in the red zone of the paper tape or a weight-for-age or height-for-age z-score of less than or equal to -3.0, the child will be excluded from the study due to malnutrition, and the parents will be advised to take the child to the nearest malnutrition clinic

Ages: 24 Months to 84 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change in executive cognitive function | Baseline and end line (12 weeks difference)
  Two measures of executive function, working memory and task-switching abilities, will be administered through play-based games by local research team members. "Spin the Pots" and "Reverse Categorization" tasks, modeled after Carlson et al., have been age modified and culturally adopted.

SECONDARY OUTCOMES:
Supplementation Attendance | Through study completion (12 weeks)
  community health workers will record attendance of children to consume the supplement.
Sicknesses | Through study completion (12 weeks)
  Community health workers will record sickness (malaria, stomach issues, fever) if children to consume the supplement are unwell.
Change in hand grip strength | Baseline and end line (12 weeks difference)
  . In the children aged 6-6.5 years, grip strength in both hands will be measured in duplicate using a dynamometer suitable for pediatric populations
Change in Hemoglobin | Baseline and end line (12 weeks difference)
  Hemoglobin will be measured non-invasively using a standard technique that uses light of different wavelengths directed at the finger
Change in skin carotenoids | Baseline and end line (12 weeks difference)
  a non-invasive optical measure of carotenoids in tissue, measured by shining light in the palm of the hand
Change in immune function | Baseline and end line (12 weeks difference)
  In this study we will measure delayed-type hypersensitivity (DTH) response using a standard Mantoux test composed of 3 antigens and a negative control via 4 intradermal skin injections that will be performed at baseline and the end of the study
Food Product Acceptability | Baseline
  Mothers (for the young children) and school children will be asked on a 4-point scale of '1=not at all' '2=a little', '3=moderately' and '4=very much' how much they enjoy eating the two types biscuits and the multivitamin. Preference for one biscuit over another will be determined by a higher total summed up score. The biscuit with a greater score will be used during the study.
Mother's Height Change | Baseline and end line (12 weeks difference)
  Height of the mothers measured in cm.
Mother's Weight Change | Baseline and end line (12 weeks difference)
  Weight of the mothers measured in kg.
Mother's MUAC change | Baseline and end line (12 weeks difference)
  The weight, height and MUAC of the mothers will also be measured, and family demographic data (family size, number of wives and children and ages) will be collected by questioning the mother.
Family Demographics Change | Baseline and end line (12 weeks difference)
  Family demographic data (family size, number of wives and children and ages) will be collected by questioning the mother.
Photographs | through study completion, 12 weeks
  Parents (and children, in the case of the school children) will be asked for permission to take photographs of them that illustrate the outcome measurements and supplement consumption, for the purpose of using in presentations on the research.
Change in weight | Baseline and end line (12 weeks difference)
  Multiple measurements of weight to ±0.1 kg will be taken using a calibrated digital scale
Change in height | Baseline and end line (12 weeks difference)
  Duplicate measures of height will be made with an upright stadiometer measuring to 0.1 cm
Change in circumferences | Baseline and end line (12 weeks difference)
  Duplicate measurements of mid-upper arm circumference (MUAC) will be taken at the midpoint between the acromion process of scapula and olecranon process, and head circumference will be measured in duplicate at the widest diameter, using standardized World Health Organization (WHO) methods.
Brain Hemoglobin | Endline at up to 12 weeks
  Near infrared spectroscopy
Brain Oxygenation | Endline at up to 12 weeks
  Near infrared spectroscopy
Brain Blood Flow | Endline at up to 12 weeks
  Near infrared spectroscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Jean Mayer USDA Human Nutrition Research Center on Aging at Tufts University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes